CLINICAL TRIAL: NCT02964182
Title: Evaluating Concomitant Use of Very Low Nicotine Content Cigarettes and E-Cigarettes Among Daily and Non-Daily Smokers
Brief Title: Very Low Nicotine Content Cigarettes and E-Cigarettes in Promoting Smoking Cessation in Daily and Intermittent Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-0638; NCI-2019-02501 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0638 (Other: M D Anderson Cancer Center); National Cancer Institute; R01DA042526 (NIH)
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Cigarette Smoking-Related Carcinoma; Tobacco-Related Carcinoma
MeSH Terms: interventions — Tobacco Products; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (usual cigarettes, VLNCC, ECIG-Hi, ECIG-Lo) (Experimental): PHASE I: Patients smoke their usual cigarettes brand during week 1.
  PHASE II: Patients smoke VLNCC cigarettes provided during weeks 2-4.
  PHASES III-IV: Patients smoke ECIG-Hi for 3 weeks and then ECIG-Lo for 3 weeks.
  Interventions: Drug: Cigarette; Drug: Nicotine Replacement; Other: Questionnaire Administration; Other: Survey Administration; Drug: Very Low Nicotine Content Cigarette; Device: ECIG-Hi; Device: ECIG-Lo
- Arm II (usual cigarettes, VLNCC, ECIG-Hi, ECIG-Lo) (Experimental): PHASE I: Patients smoke their usual cigarettes brand during week 1.
  PHASE II: Patients smoke VLNCC cigarettes provided during weeks 2-4.
  PHASES III-IV: Patients smoke ECIG-Lo for 3 weeks and then ECIG-Hi for 3 weeks.
  Interventions: Drug: Cigarette; Drug: Nicotine Replacement; Other: Questionnaire Administration; Other: Survey Administration; Drug: Very Low Nicotine Content Cigarette; Device: ECIG-Hi; Device: ECIG-Lo

INTERVENTIONS:
Drug: Cigarette — Smoke usual brand of cigarettes
Drug: Nicotine Replacement — Received NRT (Electronic Cigarette - ECIG-Hi)
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Arm I (usual cigarettes, VLNCC, ECIG-Hi, ECIG-Lo)
Drug: Nicotine Replacement — Received NRT (Electronic Cigarette - ECIG-Hi)
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Arm II (usual cigarettes, VLNCC, ECIG-Hi, ECIG-Lo)
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Drug: Very Low Nicotine Content Cigarette — Smoke very low nicotine content cigarette
  Other Names: VLNCC
Device: ECIG-Hi — Patients smoke ECIG-Hi for 3 weeks and then ECIG-Lo for 3 weeks.
Device: ECIG-Lo — Patients smoke ECIG-Lo for 3 weeks and then ECIG-Hi for 3 weeks

SUMMARY:
This trial studies what would happen if the nicotine levels in cigarettes are greatly reduced, but electronic cigarettes containing different amount of nicotine are available. Different levels of nicotine may effect certain behaviors, including withdrawal symptoms, nicotine cravings, and mood and may lead to changes in smoking behavior in current daily and intermittent smokers..

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the effects of switching to VLNCCs plus ECIG-Hi or ECIG-Lo nicotine doses on abuse liability among daily and intermittent smokers.

EXPLORATORY OBJECTIVES:

I. To explore the effects of switching to VLNCCs plus ECIG-Hi or ECIG-Lo nicotine doses on abuse liability using biochemical measures of product use, compensation, and toxicant exposure, and self-reported measures of withdrawal, craving, affect, and satisfaction.

II. To explore the effects of switching from usual-brand cigarettes to VLNCCs, and from VLNCCs to VLNCC+ECIGs on measures of abuse liability.

III. To characterize the effects of dual use of VLNCC and JUUL ECIGs on abuse liability.

OUTLINE:

PHASE I: Patients smoke their usual cigarettes brand during week 1.

PHASE II: Patients smoke VLNCC cigarettes provided during weeks 2-4.

PHASES III-IV: Patients are randomized to 1 of 2 arms.

ARM I: Patients smoke ECIG-high (Hi) for 3 weeks and then ECIG-low (Lo) for 3 weeks

ARM II: Patients smoke ECIG-Lo for 3 weeks and then ECIG-Hi for 3 weeks.

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Sign consent and agree to all study procedures
* Have an address where he/she can receive mail
* Have a device available to conduct telehealth visit (e.g., smartphone, computer, tablet, internet access, etc.)
* Able to follow verbal and written instructions in English
* Willing and able to complete two spirometry sessions (this criterion waived during COVID-19 pandemic)
* Be the only participant in their household
* Interested in trying novel nicotine products
* Daily smokers: >= 1 cigarette/little cigar per day
* Intermittent smokers: >= 1 cigarette/little cigar per day 4 to 27 days per month
* Agrees to comply with all MD Anderson institutional policies related to COVID-19 screening prior to each in-person research visit
* The individual agrees to not engage in study procedures or interactions with study personnel while operating a vehicle

Exclusion Criteria:

* Unwilling to refrain from other e-cigarette use for the duration of the study, other than what is provided to them for study purposes
* Current/recent use of certain medications:

  * Smoking cessation meds (past 90 days; e.g., wellbutrin, bupropion, Zyban, nicotine replacement therapy [NRT], Chantix)
  * Certain medications to treat depression (last 14 days; e.g., amitriptyline)
  * A case by case determination will be made by study physician for medication on the precautionary list, (e.g. nitroglycerin)
  * Self-reported daily use of opioids for 30 days or more on phone screen or at screening is exclusionary however pro re nata (PRN) use is allowed (e.g., 3 to 7 days per week or less or if more frequent, use less than a month's duration
* Unstable medical condition as determined by the medical team
* Self-reported bronchial or respiratory infection in the last 14 days (this criterion waived during COVID-19 pandemic)
* Subject's spirometry forced expiratory volume in 1 second (FEV1) percentage reading is < 50 (severe to very severe obstruction) (this criterion waived during COVID-19 pandemic)
* Self-reported abnormal heart rhythms or cardiovascular disease (stroke, chest pain, heart attack) in the last 3 months
* Meet criteria for major depressive syndrome or suicidality on the Patient Health Questionnaire-9 (PHQ-9)
* Self report of past or current diagnosis of bi-polar disorder or schizophrenia/schizoaffective disorder
* Self-reported other tobacco use besides cigarettes or little cigars (e.g., hookah, cigarillos, smokeless tobacco, chewing tobacco, pipes, cigars, etc.) on 10 or more days in the last month
* Recent (past 90 days), current, or planned (within the next 45 days) involvement in smoking cessation activities
* Positive urine pregnancy test at screening. Women who are two years post-menopausal, or who have had a tubal ligation or a partial or full hysterectomy will not be subject to a urine pregnancy test
* Women that are breastfeeding or of childbearing potential and not protected by a medically acceptable, effective method of birth control while enrolled in the study. Medically acceptable contraceptives include:

  * Approved hormonal contraceptives (such as birth control pills, patches, implants or injections)
  * Barrier methods (such as condom or diaphragm) used with a spermicide, or
  * An intrauterine device (IUD)
  * Contraceptives sold for emergency use after unprotected sex are not acceptable methods for routine use
* Subject considered by the investigator to be unsuitable to participate in the study (e.g., due to cognitive deficits or instability to last the entire duration of the study)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cinciripini, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were adults residing in the Houston metropolitan area
Pre-assignment Details: Overall, 1129 individuals were screened for interest and eligibility. Of those screened, 461 were ineligible and 455 declined to participate. A total of 213 participants were randomized.
Groups:
- Phase 1: Usual Brand Cigarette Phase (eGo Arm); Phase 1: Usual Brand Cigarette Phase (JUUL Arm): One week of smoking usual brand cigarettes
- Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm); Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm): Three weeks of smoking very low nicotine content cigarette (VLNCC)
- Phase 3 VLNCCs + Low-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + High-dose ECs (eGo Arm): Three weeks (Phase 3) of smoking very low nicotine content cigarettes (VLNCCs) and using eGo-brand low-dose electronic cigarettes (8 mg/ml freebase nicotine), followed by three weeks (Phase 4) of smoking VLNCCs and using eGo-brand high-dose electronic cigarettes (36 mg/ml freebase nicotine)
- Phase 3 VLNCCs + High-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + Low-dose ECs (eGo Arm): Three weeks (Phase 3) of smoking very low nicotine content cigarettes (VLNCCs) and using eGo-brand high-dose electronic cigarettes (36 mg/ml freebase nicotine), followed by three weeks (Phase 4) of smoking VLNCCs and using eGo-brand low-dose electronic cigarettes (8 mg/ml freebase nicotine)
- Phase 3 VLNCCs + Low-dose ECs, Then Phase 4 VLNCCs + High-dose ECs (JUUL Arm): Three weeks (Phase 3) of smoking very low nicotine content cigarettes (VLNCCs) and using JUUL-brand low-dose electronic cigarettes (3%; 35 mg/ml protonated nicotine), followed by three weeks (Phase 4) of smoking VLNCCs and using JUUL-brand high-dose electronic cigarettes (5%; 59 mg/ml protonated nicotine)
- Phase 3 VLNCCs + High-dose ECs, Then Phase 4 VLNCCs + Low-dose ECs (JUUL Arm): Three weeks (Phase 3) of smoking very low nicotine content cigarettes (VLNCCs) and using JUUL-brand high-dose electronic cigarettes (5%; 59 mg/ml protonated nicotine), followed by three weeks (Phase 4) of smoking VLNCCs and using JUUL-brand low-dose electronic cigarettes (3%; 35 mg/ml protonated nicotine)
Period: Phase 1 (Week 1)
Arm/Group | Phase 1: Usual Brand Cigarette Phase (eGo Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | Phase 3 VLNCCs + Low-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + High-dose ECs (eGo Arm) | Phase 3 VLNCCs + High-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + Low-dose ECs (eGo Arm) | Phase 1: Usual Brand Cigarette Phase (JUUL Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | Phase 3 VLNCCs + Low-dose ECs, Then Phase 4 VLNCCs + High-dose ECs (JUUL Arm) | Phase 3 VLNCCs + High-dose ECs, Then Phase 4 VLNCCs + Low-dose ECs (JUUL Arm)
Started | 176 | 0 | 0 | 0 | 37 | 0 | 0 | 0
Completed | 176 | 0 | 0 | 0 | 37 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Weeks 2-4)
Arm/Group | Phase 1: Usual Brand Cigarette Phase (eGo Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | Phase 3 VLNCCs + Low-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + High-dose ECs (eGo Arm) | Phase 3 VLNCCs + High-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + Low-dose ECs (eGo Arm) | Phase 1: Usual Brand Cigarette Phase (JUUL Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | Phase 3 VLNCCs + Low-dose ECs, Then Phase 4 VLNCCs + High-dose ECs (JUUL Arm) | Phase 3 VLNCCs + High-dose ECs, Then Phase 4 VLNCCs + Low-dose ECs (JUUL Arm)
Started | 0 | 176 | 0 | 0 | 0 | 37 | 0 | 0
Completed | 0 | 158 | 0 | 0 | 0 | 22 | 0 | 0
Not Completed | 0 | 18 | 0 | 0 | 0 | 15 | 0 | 0
Not completed — Lost to Follow-up | 0 | 7 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 11 | 0 | 0 | 0 | 1 | 0 | 0
Period: Phase 3 (Weeks 5-7)
Arm/Group | Phase 1: Usual Brand Cigarette Phase (eGo Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | Phase 3 VLNCCs + Low-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + High-dose ECs (eGo Arm) | Phase 3 VLNCCs + High-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + Low-dose ECs (eGo Arm) | Phase 1: Usual Brand Cigarette Phase (JUUL Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | Phase 3 VLNCCs + Low-dose ECs, Then Phase 4 VLNCCs + High-dose ECs (JUUL Arm) | Phase 3 VLNCCs + High-dose ECs, Then Phase 4 VLNCCs + Low-dose ECs (JUUL Arm)
Started | 0 | 0 | 78 | 80 | 0 | 0 | 10 | 12
Completed | 0 | 0 | 72 | 73 | 0 | 0 | 9 | 9
Not Completed | 0 | 0 | 6 | 7 | 0 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 3
Period: Phase 4 (Weeks 8-10)
Arm/Group | Phase 1: Usual Brand Cigarette Phase (eGo Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | Phase 3 VLNCCs + Low-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + High-dose ECs (eGo Arm) | Phase 3 VLNCCs + High-dose Electronic Cigarettes (ECs), Then Phase 4 VLNCCs + Low-dose ECs (eGo Arm) | Phase 1: Usual Brand Cigarette Phase (JUUL Arm) | Phase 2: Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | Phase 3 VLNCCs + Low-dose ECs, Then Phase 4 VLNCCs + High-dose ECs (JUUL Arm) | Phase 3 VLNCCs + High-dose ECs, Then Phase 4 VLNCCs + Low-dose ECs (JUUL Arm)
Started | 0 | 0 | 72 | 73 | 0 | 0 | 9 | 9
Completed | 0 | 0 | 68 | 70 | 0 | 0 | 8 | 9
Not Completed | 0 | 0 | 4 | 3 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- eGo Arm: Participants enrolled in the eGo Arm of this crossover design trial
- JUUL Arm: Participants enrolled in the JUUL Arm of this crossover design trial
- Total: Total of all reporting groups
Arm/Group | eGo Arm | JUUL Arm | Total
Number analyzed (Participants) | 176 | 37 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.34 (11.95) | 43.65 (11.28) | 41.74 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 16 | 96
  Male | 96 | 21 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 2 | 19
  Not Hispanic or Latino | 159 | 35 | 194
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 77 | 11 | 88
  White | 75 | 20 | 95
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 19 | 2 | 21
Region of Enrollment [Number; unit: participants]
  United States | 176 | 37 | 213

OUTCOME MEASURES:

1. Primary Outcome: Usual Brand Cigarettes Per Day
Description: Mean usual brand cigarettes per day (CPD) smoked during the phase
Time Frame: One to three weeks
Measure: Least Squares Mean (Standard Error); unit: Cigarettes per Day
Groups:
- Usual Brand Cigarette Phase (eGo Arm); Usual Brand Cigarette Phase (JUUL Arm): One week of smoking usual brand cigarettes
- Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm); Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm): Three weeks of smoking very low nicotine content cigarette (VLNCC)
- VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm): Three weeks of smoking very low nicotine content cigarettes (VLNCCs) and using eGo-brand low-dose electronic cigarettes (8 mg/ml freebase nicotine)
- VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm): Three weeks of smoking very low nicotine content cigarettes (VLNCCs) and using eGo-brand high-dose electronic cigarettes (36 mg/ml freebase nicotine)
- VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm): Three weeks of smoking very low nicotine content cigarettes (VLNCCs) and using JUUL-brand low-dose electronic cigarettes (3%; 35 mg/ml protonated nicotine)
- VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm): Three weeks (Phase 3) of smoking very low nicotine content cigarettes (VLNCCs) and using JUUL-brand high-dose electronic cigarettes (5%; 59 mg/ml protonated nicotine)
Arm/Group | Usual Brand Cigarette Phase (eGo Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm) | Usual Brand Cigarette Phase (JUUL Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm)
Number analyzed (Participants) | 176 | 168 | 146 | 149 | 37 | 36 | 18 | 21
Cigarettes per Day | 15.803 (0.5304) | 2.1563 (0.5427) | 1.8353 (0.5807) | 1.4931 (0.5751) | 12.6171 (0.9155) | 2.6665 (0.9258) | 2.3042 (1.219) | 2.1429 (1.146)

2. Primary Outcome: Very Low Nicotine Content Cigarettes Per Day
Description: Mean very low nicotine content cigarettes per day (CPD) smoked during the phase
Time Frame: One to three weeks
Population: Participants were not provided with very low nicotine content cigarettes during the Usual Brand Cigarette Phase (Phase 1)
Measure: Least Squares Mean (Standard Error); unit: Cigarettes per Day
Arm/Group | Usual Brand Cigarette Phase (eGo Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm) | Usual Brand Cigarette Phase (JUUL Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm)
Number analyzed (Participants) | 0 | 167 | 146 | 149 | 0 | 36 | 17 | 21
Cigarettes per Day |  | 15.7421 (0.9071) | 10.2652 (0.932) | 10.5811 (0.9285) |  | 12.8014 (1.6928) | 6.5151 (2.0882) | 6.2979 (1.9709)

3. Primary Outcome: Total Nicotine Equivalents (TNE)
Description: Geometric means of the natural log of total nicotine equivalents (TNE), calculated as the sum of total nicotine, total cotinine, total 3'-hydroxycotinine and nicotine N-oxide excreted in urine
Time Frame: One to three weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ln(nmol/mL)
Arm/Group | Usual Brand Cigarette Phase (eGo Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm) | Usual Brand Cigarette Phase (JUUL Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm)
Number analyzed (Participants) | 175 | 156 | 144 | 140 | 37 | 21 | 19 | 20
ln(nmol/mL) | 25.621411 [19.559 to 33.5628] | 5.37663 [3.775 to 7.6578] | 8.418756 [5.5973 to 12.6625] | 11.388661 [8.1578 to 15.899] | 35.052048 [22.5231 to 54.5506] | 5.414214 [1.8475 to 15.867] | 23.83952 [10.069 to 56.4426] | 32.428008 [13.9272 to 75.5053]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Usual Brand Cigarette Phase (eGo Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm) | Usual Brand Cigarette Phase (JUUL Arm) | Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) | VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm) | VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm)
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/176 | 0/151 | 0/152 | 0/37 | 0/37 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/176 | 3/176 | 1/151 | 0/152 | 0/37 | 0/37 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 16/176 | 52/176 | 23/151 | 18/152 | 2/37 | 1/37 | 1/19 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Brand Cigarette Phase (eGo Arm) (N=176) | Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) (N=176) | VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm) (N=151) | VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm) (N=152) | Usual Brand Cigarette Phase (JUUL Arm) (N=37) | Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) (N=37) | VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm) (N=19) | VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm) (N=21)
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Brand Cigarette Phase (eGo Arm) (N=176) | Very Low Nicotine Content Cigarette (VLNCC) Phase (eGo Arm) (N=176) | VLNCCs + Low-dose Electronic Cigarettes Phase (eGo Arm) (N=151) | VLNCCs + High-dose Electronic Cigarettes Phase (eGo Arm) (N=152) | Usual Brand Cigarette Phase (JUUL Arm) (N=37) | Very Low Nicotine Content Cigarette (VLNCC) Phase (JUUL Arm) (N=37) | VLNCCs + Low-dose Electronic Cigarettes Phase (JUUL Arm) (N=19) | VLNCCs + High-dose Electronic Cigarettes Phase (JUUL Arm) (N=21)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic Rhinitis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Appetite Decreased (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain - Cardiac (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Edema Limbs (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Elevated Co Reading (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Flu Like Symptoms (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General Disorders And Administration Site Conditions - Other, Specify (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury, Poisioning, And Procedural Complications Other (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kidney Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle Contractions (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Panic Attack (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric Disorders - Other, Specify (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Stomach Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Surgical And Medical Procedures - Other, Specify (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02964182/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT02964182/ICF_000.pdf